CLINICAL TRIAL: NCT02734914
Title: Safety and Efficacy of Suctioning Flexible Ureteroscopy With Automatic Control of Renal Pelvic Pressure : A Clinical Randomized,Controlled Study
Brief Title: Suctioning Flexible Ureteroscopy With Intelligent Control of Renal Pelvic Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Ganzhou Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Leming Song, professor, The Affiliated Ganzhou Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GanzhouHNU
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Renal Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SF-URS with automatic control of RPP (Experimental): Participants in SF-URS with automatic control of renal pelvic pressure (RPP) group undergo ureteroscopy using the intelligent pressure control device (Medical irrigation and suctioning platform with pressure feedback function, and suctioning ureteral access sheath with function of pressure measuring).
  Interventions: Device: SF-URS with automatic control of RPP
- conventional F-URS (Active Comparator): Participants in conventional F-URS group undergo ureteroscopy using the classic flexible ureteroscope.
  Interventions: Device: conventional F-URS

INTERVENTIONS:
Device: SF-URS with automatic control of RPP — A new F-URS monitoring and control of RPP using intelligent pressure control device
  Arms: SF-URS with automatic control of RPP
Device: conventional F-URS — Ureteroscopy will be conducted using the ureteral access sheath from Cook Medical to treat renal calculi.
  Arms: conventional F-URS

SUMMARY:
This study evaluates the safety and efficacy of the suctioning flexible ureteroscopy(SF-URS) with automatic control of renal pelvic pressure for the treatment of upper urinary calculi using a prospective, randomized design. Half of participants will receive suctioning flexible ureteroscopy with automatic control of renal pelvic pressure, while the other half participants will receive retrograde intrarenal surgery using the classic flexible ureteroscopy.

DETAILED DESCRIPTION:
Retrograde intrarenal surgery using flexible ureteroscope has become the first-line treatment for renal calculi < 3.0 cm and is recommended by the European Association of Urology due to its minimally-invasive nature and satisfactory result.

However, high perfusion rate leads to renal pelvic pressure increase, resulting in absorption of liquid, bacteria, and endotoxin into blood, followed by short-term complications such as systemic inflammatory response syndrome(SIRS , 8.1%), sepsis (0-4.5%), renal pelvic and ureteral tumor spread, and long-term complication of renal function impairment. Currently the commonly used flexible ureteroscope sheath (ureteral access sheath, UAS) reduces the renal pelvic pressure to a certain extent, but still can not control and monitor the renal pelvic pressure to reduce the incidence of complications, which, limit the clinical application of ureteroscopy.

Recently, the investigators present a novel technique of SF-URS with automatic control of renal pelvic pressure. In this study, transverse comparison is designed to evaluate the safety and efficacy of the suctioning flexible ureteroscopy with automatic control of renal pelvic pressure for the treatment of renal calculi.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent and indicated a willingness to comply with study treatments
* Subject has a diagnosis of renal stones according to computer tomography (CT) results
* Subject is 18-75 yrs of age
* Subject has a single stone < 3 cm in size, or multiple stones < 3 cm in cumulative size
* Subject has a serum creatinine level within the normal range for the study center

Exclusion Criteria:

* The patient who do not agree with the intention of the clinical study.
* Subject needs bilateral procedures within one-stage ureteroscopy
* Subject has an active urinary tract infection (e.g., cystitis, prostatitis, urethritis, etc.) and severe hematuria
* Subject has been diagnosed with a urethral stricture or bladder neck contracture
* Subject has a disorder of the coagulation cascade system that would put the subject at risk for intraoperative or postoperative bleeding
* Subject is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 d)
* Subject has other diseases and could not tolerate the endoscopic surgery
* Subject has any kind of anatomic abnormality of the urinary system that might have an influence on the surgery
* Subject has been diagnosed with hydronephrosis larger than 3 cm according to the B-scan ultrasonography examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
stone-free rate | 4 weeks post-operatively
  Number of participants undergo novel or conventional F-URS surgeries without residual calculus/Total number of participants in each group *100%

SECONDARY OUTCOMES:
stone-free rate | One day post-operatively
  Number of participants undergo novel or conventional F-URS surgeries without residual calculus/Total number of participants in each group *100%
Complication rates | Within 4 weeks after surgery
  Number of participants undergo novel or conventional F-URS surgeries suffer complications associated with the surgery (i.e. pain(NRS≥4), hematuria, T≥38℃, serum white blood cell≥12×〖10〗^9/L ,serum white blood cell<4×〖10〗^9/L, perforation, etc.)/Total number of participants in each group *100%

IPD SHARING:
Plan to Share IPD: Yes